CLINICAL TRIAL: NCT02913053
Title: The Effects of an Extensive Exercise Program on the Progression of Mild Cognitive Impairment (MCI)
Brief Title: The Effects of an Extensive Exercise Program on the Progression of Mild Cognitive Impairment
Acronym: NeuroExercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: German Sport University, Cologne (Other); University of Dublin, Trinity College (Other); University of Bonn (Other); University Hospital, Bonn (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZonMw733051044; BMBF 01ED1510A (Other Grant/Funding Number: German Sport University); JPND-2014-1 (Other Grant/Funding Number: Trinity College Dublin)
Record Dates: First submitted 2016-08-17; First posted 2016-09-23 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aerobic exercise (Active Comparator)
  Interventions: Behavioral: Aerobic exercise
- Stretching and Toning (Active Comparator)
  Interventions: Behavioral: Non-aerobic exercise
- Usual care: Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Aerobic exercise — Patients with mild cognitive impairment will undergo a one-year aerobic exercise program of 3 units of 45 min / week
  Arms: Aerobic exercise
Behavioral: Non-aerobic exercise — Patients with mild cognitive impairment will undergo a one-year stretching and toning (non-aerobic) exercise program of 3 units of 45 min / week
  Arms: Stretching and Toning

SUMMARY:
Exercise interventions to prevent dementia and delay cognitive decline have gained considerable attention in recent years. Human and animal studies have demonstrated that regular physical activity targets brain function by increasing cognitive reserve. Although initial studies indicate enhanced cognitive performance in patients with mild cognitive impairment (MCI) following an exercise intervention, little is known about the effect of an extensive, controlled and regular exercise regimen on the neuropathology of patients with MCI.

The aim of this study is to compare a 12- month aerobic exercise programme versus a stretching and toning (non-aerobic) programme versus a control group on the progression of cognitive decline in MCI.

It is hypothesized that MCI-related decreases in cognitive and psychomotor functioning will show less progression or even be improved after a one-year aerobic exercise intervention compared to a group of patients undergoing stretching and toning exercise as well as to a control group provided with no intervention.

DETAILED DESCRIPTION:
This randomised controlled clinical intervention study will take place across three European sites; the German Sport University Cologne, Germany, University of Nijmegen, The Netherlands and Trinity College Dublin, Ireland. Seventy-five previously sedentary patients with a clinical diagnosis of MCI will be recruited at each site. Participants will be randomised to one of three intervention arms. One group will receive a standardised one-year extensive aerobic exercise intervention (3 units of 45min / week). The second group will complete stretching and toning (non-aerobic) exercise (3 units of 45min / week) and the third group will receive usual care. Change in all outcomes will be measured at baseline (T0), after six months (T1) and after 12 months (T2).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild cognitive impairment (MCI) due to Alzheimer's disease (AD) according to the Albert et al (2011) criteria
* Montreal Cognitive Assessment (MoCA) (Nasreddine et al. 2005) score 18-26
* Stable medical condition for more than 6 months
* Stable medications for more than 3 months
* Adequate visual and auditory acuity to complete neuropsychological testin
* Electrocardiogram without significant abnormalities that might interfere with the study
* Physical ability sufficient to allow performance of endurance exercise training
* Capacity to provide written and dated informed consent form
* Medical clearance to undergo a symptom-limited cardiopulmonary exercise test and extensive aerobic exercise training
* Participants recruited from the community via newspaper articles and community advertisement will complete additional testing to determine MCI status. Participants must score ≤1.5 standard deviation (SD) of cut-off scores on episodic memory test

Exclusion Criteria:

* Diagnosis of AD or other type of dementia
* History of familial early-onset dementia
* Enrollment onto any investigational drug study
* History in the past 2 years of epileptic seizures (Participants with epilepsy who have been stable off medication and seizure free for 2 years may be included)
* Any major psychiatric disorder (a clinical diagnosis of major depressive disorder, bipolar or schizophrenia)
* Past history or MRI evidence of brain damage, including significant trauma, stroke, hydrocephalus, mental retardation, or serious neurological disorder
* Carotid stent or severe stenosis
* History of myocardial infarction within previous year congestive heart failure (New York Heart Association Class II, III or IV)
* Uncontrolled hypertension or hypotension (systolic blood pressure >200 mm Hg and/or diastolic blood pressure >110 mm Hg at rest)
* Unstable cardiac, renal, lung, liver, or other severe chronic disease
* Type 2 diabetes mellitus with hypoglycemia in the last 3 months
* Significant history of alcoholism or drug abuse within last 10 years
* Significant obesity limiting active participation in the exercise program
* Engagement in moderate-intensity aerobic exercise training for more than 30 minutes, 3 times per week, during past 2 years
* History of vitamin B12 deficiency or hypothyroidism (stable treatment for at least 3 months is allowed)
* Serious or non-healing wound, ulcer, or bone fracture

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2015-06; Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | One year
  Cognitive performance will be assessed by an extensive neuropsychological test battery

SECONDARY OUTCOMES:
Global cognitive function | One year
  MoCA (Montreal Cognitive Assessment)
Cardiovascular fitness | One year
  (sub)maximal ergometer exercise test
Physical activity | One year
  Activity monitoring with accelerometers
Health related Quality of Life | One year
  Health Related Quality of Life for People with Dementia (DemQOL)
Depressive symptoms | One year
  Center for Epidemiologic Studies Depression (CES-D)
Neuroticism-Extraversion-Openness-Five Factor Inventory (NEO-FFI) | One year
  Personality traits assessment
Timed up and Go (TUG) | One year
  Frailty measurement
Hand grip strength | One year
  Frailty measurement
30 second chair stand | One year
  Frailty measurement
Epigenetics | One year
  Genotyping of the Apolipoprotein E (APOE) 4 allele in venous blood.
Brain imaging | 6 months
  Magnetic Resonance Imaging (MRI) scan: brain structure

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schneider, Prof, Principal Investigator — German Sport University, Germany; Brian Lawlor, Prof, Principal Investigator — Trinity College Dublin, Ireland; Marcel Olde Rikkert, Prof, Principal Investigator — Radboud University, Netherlands
Locations (3):
- German Sport University, Cologne, Germany
- Trinity College Dublin, Dublin, Ireland
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stuckenschneider T, Sanders ML, Devenney KE, Aaronson JA, Abeln V, Claassen JAHR, Guinan E, Lawlor B, Meeusen R, Montag C, Olde Rikkert MGM, Polidori MC, Reuter M, Schulz RJ, Vogt T, Weber B, Kessels RPC, Schneider S. NeuroExercise: The Effect of a 12-Month Exercise Intervention on Cognition in Mild Cognitive Impairment-A Multicenter Randomized Controlled Trial. Front Aging Neurosci. 2021 Jan 14;12:621947. doi: 10.3389/fnagi.2020.621947. eCollection 2020. PMID 33519425
- [Derived] Devenney KE, Sanders ML, Lawlor B, Olde Rikkert MGM, Schneider S; NeuroExercise Study Group. The effects of an extensive exercise programme on the progression of Mild Cognitive Impairment (MCI): study protocol for a randomised controlled trial. BMC Geriatr. 2017 Mar 22;17(1):75. doi: 10.1186/s12877-017-0457-9. PMID 28330458